CLINICAL TRIAL: NCT04877314
Title: The Effect of Intermittent Fasting on Immune System
Brief Title: The Immun Status Changes Due to Intermittent Fasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof. MD, Istanbul Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Intermittent fasting immune
Record Dates: First submitted 2021-05-05; First posted 2021-05-07 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Intermittent Fasting
Keywords: Cytokine; Intermittent fasting
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Cytokine levels before and after intermittent fasting period for 3 weeks
Masking Description: Measuring the level of IL1, IL6, TNFα, IL10 cytokines before and after the 3 weeks intermittent fasting period for 30 overweight volunteers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermittent fasting (Experimental)
  Interventions: Other: Intermittent fasting

INTERVENTIONS:
Other: Intermittent fasting — 30 overweight male volunteers who will have 3 weeks intermittent fasting which has 16 hours fasting and 8 hours eating in a day period.

SUMMARY:
Positive effects of calorie restriction on quality of life and diseases are reported. Intermittent fasting, one of the calorie restriction methods, has been shown to be beneficial for health with many metabolic effects, not just calorie restriction. Preclinical studies show the disease-modifying effects of intermittent fasting in animal models on a wide variety of chronic disorders, including obesity, diabetes, cardiovascular disease, cancers, and neurodegenerative brain diseases. There are very few studies evaluating the effects of intermittent fasting on the immune system, and only TNFα, IL6 and IL10 cytokines were evaluated in these studies to evaluate the immune system. In this study, we aimed to evaluate the conditions of inflammatory markers in peripheral blood before and after intermittent fasting period in overweight volunteers with a Body Mass Index between 25 and 30. Volunteers will have intermittent fasting for 3 weeks, which conforms to the 16-hour fasting and 8-hour meal format.

DETAILED DESCRIPTION:
In a 1997 article by Weindruch and Sohal, they reported that reducing food availability (calorie restriction) throughout life has significant effects on aging and lifespan in animals. There are many modalities for calorie restriction, one of which is intermittent fasting. Intermittent fasting involves having little or no energy intake during a certain period of the day, then free intake of energy for the rest of the day. Some of the modalities applied in this context can be listed as 12 hours fasting-12 hours eating, 16 hours fasting-8 hours eating, 20 hours fasting-4 hours eating. Studies in animals and humans show that most of the health benefits of intermittent fasting are not just the result of decreased free radical production or weight loss. Instead, intermittent fasting elicits cellular responses that can adapt to improve glucose regulation between and within organs, increase stress resistance, and suppress inflammation. During intermittent fasting, cells activate pathways that increase their defenses against oxidative and metabolic stress and remove or repair damaged molecules.Preclinical studies show the disease-modifying effects of intermittent fasting in animal models on a wide variety of chronic disorders, including obesity, diabetes, cardiovascular disease, cancers, and neurodegenerative brain diseases . Periodic opening and closing of metabolism with intermittent fasting not only provides the ketones necessary for cells to use during the fasting period, but also elicits highly regulated systemic and cellular responses to increase mental and physical performance and disease resistance.

There are very few studies evaluating the effects of intermittent fasting on the immune system, and only TNFα, IL6 and IL10 cytokines were evaluated in these studies to evaluate the immune system. In one of these studies, it was reported that proinflammatory cytokines of TNFα, IL6, which were measured after intermittent fasting for 30 days for 14 hours, decreased significantly.

In this study, the investigators aimed to evaluate the effect of 16-hour fasting and 8-hour intermittent fasting application on overweight volunteers with a Body Mass Index of 25-30 for inflammatory markers in peripheral blood .

ELIGIBILITY:
Inclusion Criteria:

* Bady mass index should be between 25-30
* Male

Exclusion Criteria:

* Diabetes patients,
* Immune deficiency history,
* Cancer patients,
* Individuals who did not agree to participate in the study

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Hormonal factors could affect cytokine values over time
Enrollment: 20 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Cytokine levels | 3 weeks
  IL1, IL6, TNFα, IL10 cytokine levels

SECONDARY OUTCOMES:
Demographic values | 3 weeks
  Weight as kilograms, Height as meters

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk O Idiz, Assoc.Prof., Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If the study complete, we could share

REFERENCES:
- [Background] Weindruch R, Sohal RS. Seminars in medicine of the Beth Israel Deaconess Medical Center. Caloric intake and aging. N Engl J Med. 1997 Oct 2;337(14):986-94. doi: 10.1056/NEJM199710023371407. No abstract available. PMID 9309105
- [Background] Panda S. Circadian physiology of metabolism. Science. 2016 Nov 25;354(6315):1008-1015. doi: 10.1126/science.aah4967. PMID 27885007
- [Background] Di Francesco A, Di Germanio C, Bernier M, de Cabo R. A time to fast. Science. 2018 Nov 16;362(6416):770-775. doi: 10.1126/science.aau2095. PMID 30442801